CLINICAL TRIAL: NCT03213119
Title: Boosting Reward-based Attention Through VEstibular STimulation
Acronym: BRAVEST
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: number of planned study inclusions not achievable
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL17_0263; 2017-A01784-49 (Other: ID-RCB)
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Brain Lesion of the Right Hemisphere; Unilateral Spatial Neglect for Half of Them
Keywords: Caloric Vestibular Stimulation Reward; Brain Stimulation; Reward; Vestibular System; Cingulate Cortex; Cancellation Tasks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caloric Vestibular Stimulation, Left-Warm (Experimental): Caloric Vestibular Stimulation (CVS) stimulates the vestibular system through thermic currents applied through small quantity of water injected in the external ear. The Left-Warm condition uses water with a temperature of 44°. It induces a nystagmus with its slow phase towards the right.
  Interventions: Procedure: Non-invasive brain stimulation of the vestibular system through caloric vestibular stimulation.
- Caloric Vestibular Stimulation, Left-Cold (Experimental): Caloric Vestibular Stimulation (CVS) stimulates the vestibular system through thermic currents applied through small quantity of water injected in the external ear. The Left-Cold condition uses water with a temperature of 30°. It induces a nystagmus with its slow phase towards the left.
  Interventions: Procedure: Non-invasive brain stimulation of the vestibular system through caloric vestibular stimulation.
- Caloric Vestibular Stimulation, SHAM (Sham Comparator): The SHAM condition uses water with a temperature of 37°. It does not induce nystagmus
  Interventions: Procedure: Non-invasive brain stimulation of the vestibular system through caloric vestibular stimulation.

INTERVENTIONS:
Procedure: Non-invasive brain stimulation of the vestibular system through caloric vestibular stimulation. — Caloric vestibular stimulation (CVS) involves the irrigation of cold or warm water into the external ear canal, and induces a temperature gradient across the semicircular canals stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function.
  Arms: Caloric Vestibular Stimulation, Left-Warm
Procedure: Non-invasive brain stimulation of the vestibular system through caloric vestibular stimulation. — Caloric vestibular stimulation (CVS) involves the irrigation of cold or warm water into the external ear canal, and induces a temperature gradient across the semicircular canals stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function.
  Arms: Caloric Vestibular Stimulation, Left-Cold
Procedure: Non-invasive brain stimulation of the vestibular system through caloric vestibular stimulation. — Caloric vestibular stimulation (CVS) involves the irrigation of cold or warm water into the external ear canal, and induces a temperature gradient across the semicircular canals stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function. The SHAM condition uses body-temperature water, and thus does not result into vestibular unbalance.
  Arms: Caloric Vestibular Stimulation, SHAM

SUMMARY:
The exploration of space is more effective when intrinsically rewarding elements are located in the visual scene. Thus, rewards could be exploited as a novel rehabilitation approach to various attentional disorders. The first part of the project aims to characterize these effects at the behavioural level. The interventional part consists then in the administration of Caloric Vestibular Stimulation (CVS), which by means of injection of a small quantity of water in the external ear activates the vestibular organs and subsequently vestibular-related brain areas. Among the observed brain activations, the possibility to reach cingulate areas appears particularly interesting because it foreshadows the possibility to further enhance attentional capture by rewards.

CVS will be delivered to patients with brain lesion of the right hemisphere, engaged in cancellation tasks requiring the processing of targets of different nature (e.g. monetary or neutral). The main prediction is that CVS administration would enhance spatial exploration in terms of center of gravity of the cancellation and improved accuracy as a function of the type of target processed (e.g. its value).

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age, less than 85
* right handed
* Benefit of social health security
* Normal or corrected-to-normal vision
* Brain lesion localised in the right hemisphere, confirmed by CT or MRI

Exclusion Criteria:

* Anamnesis of neurological of psychiatric illness
* Pregnancy or breastfeeding
* Administrative measures restricting legal rights
* Recent participation to other brain stimulation studies (< 1 week)
* Perforation of the tympanic membrane
* Anamnesis of recurrent otitis media

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2023-02-13 (Estimated)

PRIMARY OUTCOMES:
Center of Gravity (pixels). | Days 1, 2, and 3
  For line bisection defined as the difference between participants' mark and the objective center of the line. For cancellation tasks it is calculated as the grand average of horizontal and vertical coordinates of all the marks. In both cases smaller indices indicate a leftward exploration bias, whereas larger indices indicate rightward bias.

SECONDARY OUTCOMES:
Reaction times (ms). | Days 1, 2, and 3.
  The speed of response is a traditional indicator of the amount of cognitive processing underneath provided responses. It is measured by professional programs (e.g. Presentation) running on standard PCs
Response accuracy (%) | Days 1, 2, and 3.
  The proportion of correct responses provided, automatically computed by professional programs (e.g. Presentation) running on standard PCs.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CRNL, équipe IMPACT (CNRS UMR5292, INSERM U1028), Bron
  - Service de médecine et réadaptation neurologique, Hôpital Henry Gabrielle, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: No